CLINICAL TRIAL: NCT01856127
Title: A Randomized, Double-Blind, Active Controlled Clinical Trial of Switching to Vilazodone for Antidepressant-Associated Sexual Dysfunction
Brief Title: Does Vilazodone Help With Antidepressant-associated Sexual Dysfunction?
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: PI left institution
Sponsor: Thomas Jefferson University (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VII-IT-09; VII-IT-09 (Other Grant/Funding Number: Forest Research Institute)
Record Dates: First submitted 2013-03-21; First posted 2013-05-17 (Estimated); Last update posted 2016-08-25 (Estimated); Status verified 2016-08

CONDITIONS: Sexual Dysfunction; Major Depressive Disorder
Keywords: Sexual Dysfunction; Antidepressant; Major Depressant; SSRI; SNRI; Vilazodone; Sertraline
MeSH Terms: conditions — Sexual Dysfunction, Physiological; Depressive Disorder, Major | interventions — Vilazodone Hydrochloride; Sertraline

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vilazodone (Experimental): Vilazodone
  Interventions: Drug: Vilazodone
- Sertraline (Active Comparator): Sertraline
  Interventions: Drug: Sertraline

INTERVENTIONS:
Drug: Vilazodone — Vilazodone is a newly introduced antidepressant which, in contrast to the selective serotonin reuptake inhibitors (SSRIs) and serotonin-norepinephrine reuptake inhibitors (SNRIs) appears to have a minimal adverse effect on sexual functioning
  Other Names: Viibryd
  Arms: Vilazodone
Drug: Sertraline — Sertraline hydrochloride (trade names Zoloft, Lustral) is an antidepressant of the selective serotonin reuptake inhibitor (SSRI) class.
  Other Names: Zoloft
  Arms: Sertraline

SUMMARY:
This is a three-center, randomized, double-blind, fixed dose study designed to assess the efficacy, safety, and tolerability of a switch to vilazodone for sexual dysfunction associated with use of a selective serotonin reuptake inhibitor (SSRI) and serotonin-norepinephrine reuptake inhibitor (SNRI)compared to switching to sertraline in patients with Major Depressive Disorder (MDD).

Vilazodone is a newly introduced, FDA approved antidepressant that is a combined serotonin specific reuptake inhibitor and serotonin 1A receptor partial agonist. In contrast to the SSRIs and SNRIs, appears to have low adverse effects on sexual functioning when compared to placebo.

DETAILED DESCRIPTION:
The design will be a randomized, double blind study with patients being randomized to switching to either vilazodone or sertraline. This will consist of a 1-week Screening phase, a 2-week Cross Taper phase, an 8-week Treatment phase, and an optional 2-week Down taper phase. The total duration of each patient's participation will be 13 weeks.

Seventy-two patients will be randomized at the Baseline visit to either vilazodone or sertraline, 24 at each of the 3 sites. Patients will be recruited over 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be able to understand the nature of the study, agree to comply with the prescribed dosage regimens, report for regularly scheduled office visits, and communicate to study personnel about adverse events and concomitant medication use;
2. Patients with major depressive disorder who are being treated with a selective serotonin reuptake inhibitor (citalopram, escitalopram, fluvoxamine, or paroxetine) or serotonin-norepinephrine reuptake inhibitor (desvenlafaxine, duloxetine, venlafaxine) for a minimum of 8 weeks.
3. The current episode of MDD is in remission (MADRS score < 10 and CGI score of 1 or 2)
4. The duration of the current MDD episode is less than 2 years
5. Presence of antidepressant-associated sexual dysfunction (i.e., absence of sexual dysfunction prior to becoming depressed and presence of significant dysfunction while on the SSRI or SNRI despite being in remission from the depression).
6. Patient is at least 18 years old and not more than 65 years old
7. Patients must have the opportunity for sexual activity during the study period (in the form of availability of a suitable partner for sexual activity and/or openness to masturbation)
8. Patients must be willing to attempt some sexual activity (including masturbation) at least once every two weeks during the study

Exclusion Criteria:

1. Patients who have previously failed to respond to or to tolerate either vilazodone or sertraline.
2. Patients with a history of severe discontinuation symptoms on tapering off the current antidepressant
3. Patients with other known causes of sexual dysfunction
4. Use of prohibited medications during the study period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2013-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Changes in Sexual Functioning Questionnaire (CSFQ (c)) | Baseline-11 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rajnish Mago, MD, Principal Investigator — Thomas Jefferson University; Michael Thase, MD, Principal Investigator — University of Pennsylvania; Anita Clayton, MD, Principal Investigator — University of Virginia
Locations (3):
- United States (3):
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No